CLINICAL TRIAL: NCT05458336
Title: Saline Nasal Irrigations to Eradicate SARS-CoV-2
Brief Title: A Randomized Controlled Clinical Trial on the Use of Saline Nasal Irrigations to Eradicate Localized Nasal Infection by SARS-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 991/CE MARCA
Record Dates: First submitted 2022-06-28; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Symptoms and Signs
MeSH Terms: conditions — Signs and Symptoms | interventions — Nasal Lavage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Experimental): Subjects who have been given nasal lavages
  Interventions: Device: Nasal lavages with Tonimer Panthexyl®
- Controls (No Intervention): Subjects who haven't been given nasal lavages

INTERVENTIONS:
Device: Nasal lavages with Tonimer Panthexyl® — At the moment of diagnosis, patients were asked to fill out an ad hoc questionnaire to subjectively evaluate symptoms and comorbidities at the moment of diagnosis and of negativization. Subjects performed a daily nasal swab. When the subjects tested negative for the first time, they had to complete the questionnaire once again. Patients were given nasal washes (Tonimer Panthexyl®) to be performed three times a day, and in any case after nasal swab.
  Arms: Cases

SUMMARY:
Consecutive adult (>18 years old) subjects who tested positive for SARS-CoV-2 with nasopharyngeal swab at the local COVID-19 Prevention Centre were included.

Patients were divided into two groups: cases (who performed nasal lavages) and controls (who did not perform lavages), with similar confounding factors (age, comorbidities, vaccination status).

At the moment of diagnosis, patients were asked to fill out an ad hoc questionnaire to evaluate their symptoms at the moment of diagnosis and of negativization.

Subjects were asked to perform, at a daily time of their choice, a nasal swab provided at the moment of enrolment. When the subjects tested negative for the first time, they had to complete the questionnaire once again.

The study was divided into two phases. In the first phase cases were recruited and were given nasal washes (Tonimer Panthexyl®) to be performed three times a day, and in any case after nasal swab. In the second phase controls were recruited and were asked to perform only daily nasal swabs.

Symptoms course and time of negativization were analyzed. Statistic comparisons were made using Kaplan-Meier test. P values <0,05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* starting participation to the study within the first 48 hours since diagnosis
* ability in self-swabbing
* ability in self-administration of nasal lavages

Exclusion Criteria:

* age <18 years
* refusal of participation
* starting participation to the study after the first 48 hours since diagnosis
* no ability in self-swabbing
* no ability in self-administration of nasal lavages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Symptoms' course | From date of the first positive swab until the date of to the first negative swab, up to 14 days
  Evaluation of differences in disease's course between cases and controls by filling an ad hoc questionnaire about symptoms

SECONDARY OUTCOMES:
Time of negativization | From date of the first positive swab until the date of to the first negative swab, up to 14 days
  Evaluation of differences in negativization time between cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Spinato, MD, Study Chair — Universiry of Padova
Locations (1):
- Unit of Otorhinolaryngology of Treviso Hospital, Treviso, Italy